CLINICAL TRIAL: NCT05760534
Title: Ideal Dosage for Sedation of Obese Patients Undergoing Knee or Hip Arthroplasty Under Spinal Anesthesia - a Phase 4 Clinical Trial
Brief Title: Ideal Dosage for Sedation of Obese Patients Undergoing Knee or Hip Arthroplasty Under Spinal Anesthesia
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Seoul National University Hospital (Other)
Responsible Party: Principal Investigator, Jin-Tae Kim, Professor, Seoul National University Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: H-2301-016-1391
Record Dates: First submitted 2023-02-26; First posted 2023-03-08 (Actual); Last update posted 2025-12-29 (Actual); Status verified 2025-12

CONDITIONS: Arthritis Knee; Arthritis Hip
MeSH Terms: interventions — remimazolam

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Ideal body weight group (Experimental)
  Interventions: Drug: Remimazolam
- Total body weight group (Active Comparator)
  Interventions: Drug: Remimazolam

INTERVENTIONS:
Drug: Remimazolam — 0.075 mg/kg Remimazolam will be loaded over 1 min, then continuously infused at 0.2-1.0 mg/kg/h based on ideal or total body weight

SUMMARY:
This study aims to compare ideal body weight- and total body weight-based dosage for remimazolam sedation of obese patients undergoing knee or hip arthroplasty under spinal anesthesia.

ELIGIBILITY:
Inclusion Criteria:

* Patients scheduled for elective knee or hip arthroplasty under spinal anesthesia
* BMI>25
* American Society of Anesthesiologists (ASA) classification I, II, III

Exclusion Criteria:

* Patient refusal
* Contraindication for spinal anesthesia
* Contraindication for remimazolam infusion
* History of hypersensitivity to remimazolam
* History of chronic use of benzodiazepine or opioid
* Baseline MOAA/S score of 4 or lower
* Pregnancy

Ages: 19 Years to 79 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 110 (Actual)
Dates: Start 2023-03-06 (Actual); Primary Completion 2025-11-25 (Actual); Study Completion 2025-11-25 (Actual)

PRIMARY OUTCOMES:
Incidence of intraoperative respiratory depression | From entrance to exit from the operating room
  Incidence of intraoperative respiratory depression

SECONDARY OUTCOMES:
Total remimazolam infusion dose | From start to end of remimazolam infusion
  Total remimazolam infusion dose (mg/kg/h)
Incidence of intraoperative hypotension | From entrance to exit from the operating room
  Mean blood pressure <65 mmHg
Incidence of intraoperative hypertension | From entrance to exit from the operating room
  Systolic blood pressure >120% of baseline
Incidence of intraoperative bradycardia | From entrance to exit from the operating room
  Heart rate <45 bpm
Incidence of intraoperative tachycardia | From entrance to exit from the operating room
  Heart rate >120 bpm
Incidence of intraoperative oxygen desaturation | From entrance to exit from the operating room
  Pulse oximeter saturation (SpO2) < 93%
Incidence of intraoperative nausea or vomiting | From entrance to exit from the operating room
  Nausea or vomiting during surgery
Incidence of intraoperative hiccups | From entrance to exit from the operating room
  Hiccups during surgery
Incidence of intraoperative paradoxical movements | From entrance to exit from the operating room
  Paradoxical movements during surgery
Modified Observer's Assessment of Alertness/Sedation (MOAA/S) score | From start of remimazolam infusion until time of full alertness
  MOAA/S score assessment at 10 min intervals
Intraoperative Patient State Index (PSi) | From entrance to exit from the operating room
  Continuous monitoring of PSi with Sedline sensor
Time to reach MOAA/S score 5 after end of surgery | From end of remimazolam infusion until time of full alertness
  Time to reach MOAA/S score 5 (min)
Length of stay at the post-anesthesia care unit (PACU) | From entrance to exit from the PACU
  Length of stay at the PACU (min)
Patient satisfaction | At exit from PACU
  Numeric rating scale of 0 (not satisfied at all) to 10 (absolutely satisfied)
Intraoperative recall | At exit from PACU
  Assessment with the modified Brice questionnaire
Incidence of postoperative nausea or vomiting | From entrance to exit from the PACU
  Incidence of nausea or vomiting
Incidence of postoperative delirium | From end of surgery to third postoperative day
  Assessment with the Confusion Assessment Method (CAM)
Incidence of postoperative respiratory depression | From entrance to exit from the PACU
  Respiratory rate < 8/min or SpO2<93%
Incidence of postoperative hypotension | From entrance to exit from the PACU
  Mean blood pressure <65 mmHg
Incidence of postoperative hypertension | From entrance to exit from the PACU
  Systolic blood pressure >120% from baseline

CONTACTS AND LOCATIONS:
Overall Officials: Jin-Tae Kim, M.D., Ph.D., Principal Investigator — Seoul National University Hospital
Locations (1):
- Jin-Tae Kim, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: No